CLINICAL TRIAL: NCT06656728
Title: Clinical Validation Of A Diagnostic Cancerend24 Screening As An Aid To The Clinician For The Diagnosis Of Cancer In Healthy Subjects Attending The ICPC
Brief Title: CancerenD24 Screening as an Aid to the Clinician for the Diagnosis of Cancer
Acronym: CancerenD24
Status: Recruiting | Type: Observational
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Tel Aviv Medical Center (Other)
Responsible Party: Sponsor
Other Study IDs: 0365-24-TLV
Record Dates: First submitted 2024-10-22; First posted 2024-10-24 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Cancer; Early Detection of Cancer
Keywords: Cancer; Early detection; Venous blood sample; CancerenD24; CD24; CD11b; Malignant disease
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 36 Months
Biospecimen Retention: Samples Without DNA — Blood sample
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy subjects: Patients over the age of 40, without active cancer in the last 5 years, who come for a cancer screening (and sometimes other screenings) at the Integrated Cancer Prevention Center
  Interventions: Other: Blood-based liquid biopsy

INTERVENTIONS:
Other: Blood-based liquid biopsy — Venous blood sample will be taken from the patient as part of the routine blood tests taken as part of the work at the Medical Center

SUMMARY:
The purpose of the researchers is to test whether the CancerenD24 index, an algorithm based on the quantitative value of CD24, CD11b, clinical and laboratory characteristics, developed in the laboratory can help in the early detection of a malignant disease in a population of healthy subjects.

DETAILED DESCRIPTION:
CD24 is a protein found naturally in the body and serves as a natural regulator of the immune system, in order to prevent its uncontrolled and disproportionate reaction. It is known that in a normal state the CD24protein is almost never expressed in healthy cells with the exception of the white blood cells of the blood cells in the adult person. In contrast, cancer and even pre-cancer cells express high levels of CD24. Sometimes this expression is associated with a more violent course of the cancer. Similarly, CD11b is another protein that is expressed on the surface of white blood cells and affects the migration of white blood cells and their penetration into the tissue. In addition, CD11b plays an important role in the tumor microenvironment and cancer progression. And it is used as a prognostic marker. The role and involvement of these proteins (CD24/CD11b) in various cellular processes, led our group of researchers to hypothesize that an algorithm based on CD24and CD11b protein expression on white blood cells can help in the early diagnosis of cancer and assist doctors in diagnosing this serious disease in its early stages.

The test is intended for routine use, as an aid to doctors to identify most types of cancer in earlier stages. CancerenD24 is not affected by fasting and the time of day when the blood sample is taken.

In this study, it is expected to recruit 2000 male and female subjects, who will be recruited over a period of 36 months. The experiment does not involve any treatment. During the visit to the medical center, an experienced staff member will explain the study to the patient, and after agreeing to his participation, the patient will sign an informed consent form, as is customary. After that, the same staff member will interview the patient in order to obtain demographic data and information about risk factors. After that, a venous blood sample will be taken from the patient as part of the routine blood tests taken as part of the work at the Medical Center. For this purpose, patients over the age of 40, without active cancer in the last 5 years, who come for a cancer screening (and sometimes other screenings) at the Integrated Cancer Prevention Center and the Medical Center will be recruited.

ELIGIBILITY:
Inclusion Criteria:

1. Completion of all medical exams and questionnaires including cancer diagnoses, demographic data and other epidemiologic information
2. Willing and able to sign an informed consent
3. Age ≥40 years

Exclusion Criteria:

1. Age < 40 years
2. Pregnancy or breastfeeding
3. Any type of fever
4. Any cancer active at study entry or up to 5 years prior to study entry
5. Polyposis syndromes
6. Inflammatory bowel disease
7. Unwilling or unable to provide informed consent

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy patients who attend the Integrated Cancer Prevention Center
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2024-09-03 (Actual); Primary Completion 2024-09-04 (Actual); Study Completion 2027-09 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the CancerenD24 Screening Assay | 3 years
  To evaluate the "CancerenD24 screening assay" as an aid to physicians in diagnosing cancer in subjects aged 40 years and above

SECONDARY OUTCOMES:
Sensitivity and specificity of CancerenD24 versus the ground truth diagnosis | 3 years
  Sensitivity and specificity of CancerenD24 versus the ground truth diagnosis in subjects aged 40 years and above positive and negative predictive values of CancerenD24 versus the ground truth diagnosis in subjects aged 40 years and above
Positive and negative likelihood ratios of CancerenD24 versus the ground truth diagnosis | 3 years
  Positive and negative likelihood ratios of CancerenD24 versus the ground truth diagnosis in subjects aged 40 years and above
Sensitivity of the CancerenD24 versus any confirmed cancer | 12 months
  Sensitivity of the CancerenD24 versus any confirmed cancer during the full follow-up period of 12 months in subjects aged 40 years and above
CancerenD24 accuracy (sensitivity, specificity, PPV and NPV) measures | 3 months, 6 months, 9 months, 12 months
Time to cancer diagnosis | up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Integrated Cancer Prevention Center at the Tel Aviv Sourasky Medical Center Ichilov, Tel Aviv, Israel

IPD SHARING:
Plan to Share IPD: No